CLINICAL TRIAL: NCT05964660
Title: New 3D-echocardiography-based Motion Integration and mAnagement for subsTrate characteRisation and Stereotactic Arrhythmia radIoablation tX in Ventricular Tachycardias- the MATRIX-VT Study
Brief Title: Echocardiography-based Motion Integration and Management for Substrate Characterization and STAR Therapy in Ventricular Tachycardias
Acronym: MATRIX-VT
Status: Recruiting | Type: Observational
Sponsor: University of Luebeck (Other)
Collaborators: Institute for Robotics and Cognitive Systems, University of Luebeck, Germany (Unknown)
Responsible Party: Principal Investigator, Prof. Roland Richard Tilz, Professor Dr. med.univ., University of Luebeck
Other Study IDs: MATRIX-VT
Record Dates: First submitted 2023-07-19; First posted 2023-07-28 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Ventricular Arrythmia
Keywords: Ventricular arrhythmia; Ventricular tachycardia; Stereotactic arrhythmia radioablation; Artificial intelligence; Motion management; Motion integration
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- VT Patients: Patients with indication for catheter ablation of ventricular arrhythmia and preprocedural contrast-enhanced cardiac computed tomography for cardiac structure characterization.

SUMMARY:
Prospective, observational, single center, pilot study to analyze the feasibility of motion and structural data integration in patients with ventricular arrhythmia by means of artificial intelligence for improved arrhythmogenic substrate characterization and motion management during stereotactic arrhythmia radioablation.

DETAILED DESCRIPTION:
This is a prospective, observational, single center, pilot study. Data from preprocedural contrast-enhanced cardiac computed tomography and optically-tracked 3D transthoracic echocardiography of patients receiving catheter ablation for ventricular arrhythmia will be analyzed by means of artificial intelligence in order to better characterize the ventricular arrhythmogenic substrate and to improve the definition methods of the planning target volume during the stereotactic arrhythmia radioablation therapy by integrating the motion data into volume demarcation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Indication for catheter ablation of ventricular arrhythmias (ventricular fibrillation, ventricular tachycardia, premature ventricular contractions)
* Indication for preprocedural contrast-enhanced cardiac computed tomography for cardiac structure characterization

Exclusion Criteria:

* Platelet count < 100,000 cells/mm3
* BMI > 45 kg/m2 or < 18 kg/m2

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 20 patients with indication for catheter ablation of ventricular arrhythmia (VA) (ventricular tachycardia (VT), ventricular fibrillation (VF), premature ventricular contraction (PVC)) and for preprocedural contract-enhanced cardiac computed tomography (CT) for cardiac structure characterization will be prospectively enrolled in the study. The therapeutic approach follows the current clinical standard.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility of algorithm training to achieve improved arrhythmogenic substrate characterization | 1 month after complete data collection
  The feasibility of training the artificial intelligence-based algorithm using the preprocedural contrast-enhanced cardiac computed tomography and optically-tracked 3D transthoracic echocardiography data to better define the ventricular arrhythmogenic substrate in patients exhibiting ventricular arrhythmias.
Feasibility of algorithm training to improve the planning target volume definition for stereotactic arrhythmia radioablation therapy | 1 month after complete data collection
  The feasibility of training the artificial intelligence-based algorithm using the preprocedural contrast-enhanced cardiac computed tomography and optically-tracked 3D transthoracic echocardiography data to better define the planning target volume for stereotactic arrhythmia radioablation therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik für Rhythmologie, Lübeck, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No